CLINICAL TRIAL: NCT00817232
Title: Effectiveness of Microcurrent in the Treatment of Chronic Tennis Elbow - a Preliminary Trial
Brief Title: Effectiveness of Microcurrent for Treatment of Tennis Elbow
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Hertfordshire (Other)
Responsible Party: Leon Poltawski, University of Hertfordshire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEPEC/10/08/05
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-08

CONDITIONS: Tennis Elbow
Keywords: tennis elbow; microcurrent; tissue healing
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 (Experimental): 50 microamp amplitude
  Interventions: Device: Microcurrent (Elexoma Medic)
- Treatment 2 (Experimental): 500 microamp amplitude
  Interventions: Device: Microcurrent (Elexoma Medic)

INTERVENTIONS:
Device: Microcurrent (Elexoma Medic) — monophasic frequency modulated square wave current applied for 99 minutes daily for 21 days
  Other Names: Elexoma Medic

SUMMARY:
Tennis elbow is a relatively common musculoskeletal disorder that can cause significant pain and disability. Treatment of the disorder is not always successful, and it often recurs or becomes chronic. More effective management options are required. There is evidence that electric microcurrent can promote tissue healing and symptom resolution in various chronic hard and soft tissue disorders, but few human studies investigating its use with chronic tendon problems. It is an easily applied therapy with very few reports of side effects. It can be applied at home using a portable unit and, if it is clinically effective, may also prove more cost effective than other therapies.

A clinical trial is planned to evaluate the therapy but, in the absence of relevant published evidence, a preliminary study is required to look for a treatment effect and inform a power calculation for sample size, The study will also allow some investigation of dose-dependence, which is a key issue in many forms of electrotherapy. Finally it will enable evaluation of elements of the full trial protocol so that any weaknesses can be addressed before it begins.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of tennis elbow for at least 3 months
* clinical diagnosis of tennis elbow

Exclusion Criteria:

* significant symptom improvement in previous month
* receipt of any active treatment for the condition in the previous month
* currently under the care of another health professional for tennis elbow
* current cervical radiculopathy
* other pathology affecting distal upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Tendon pathology as indicated by sonography | baseline, 3 weeks, 6 weeks, 4 months
Patient-Rated Global Change Score | 3 weeks, 6 weeks, 4 months

SECONDARY OUTCOMES:
Pain Free Grip Strength | baseline, 3 weeks, 6 weeks, 4 months
Patient-rated Tennis Elbow Questionnaire | baseline, 3 weeks, 6 weeks, 4 months
Patient-Specific Functional Scale | baseline, 3 weeks, 6 weeks, 4 months
Adverse events | 3 weeks, 6 weeks, 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hertfordshire, Hatfield, Hertfordshire, United Kingdom

REFERENCES:
- See also: application of electrotherapy — http://www.electrotherapy.org